CLINICAL TRIAL: NCT05716594
Title: Clinical Evaluation of Enteral-extended Anti-reflux Stents for Pancreatic Pseudocyst
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Huang Yonghui, Chief Physician, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LM2022426
Record Dates: First submitted 2023-01-29; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Pancreatic Pseudocyst
MeSH Terms: conditions — Pancreatic Pseudocyst

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enteral-extended Anti-reflux Stents Group (Experimental): Patients are going to implant enteral-extended anti-reflux stents
  Interventions: Combination Product: Plant enteral-extended anti-reflux stents
- Traditional Stents Group (Active Comparator): Patients are going to implant traditional stents
  Interventions: Combination Product: Plant traditional stents

INTERVENTIONS:
Combination Product: Plant enteral-extended anti-reflux stents — Plant enteral-extended anti-reflux stents in EUS-guided drainage of pancreatic pseudocysts
  Arms: Enteral-extended Anti-reflux Stents Group
Combination Product: Plant traditional stents — Plant traditional stents in EUS-guided drainage of pancreatic pseudocysts
  Arms: Traditional Stents Group

SUMMARY:
At present, endoscopic therapy is the preferred method to solve biliary or pancreatic diseases. And EUS-guided stent implantation and drainage of pancreatic pseudocyst is the main method in Endoscopic treatment of pancreatic pseudocyst. However, blockage of stent is a problem that has puzzled endoscopists for a long time. The mechanism of stent blockage is related to the reflux of gastrointestinal contents into the stent. Although plastic stents are widely used in patients who needed drainage. However, the average free time for stent is only 77 to 126 days, leading to the need for stent replacement in most patients within 3 months. As one end of the double pigtail stent used for drainage of pancreatic pseudocyst may be located in the stomach, it may cause the stent to be blocked by the contents of the stomach. Therefore, multiple stents or additional stents or drainage tube are often needed to further strengthen the drainage.

It seems that the mechanism of stent blockage are associated with gastrointestinal contents reflux. And stents required be replaced again by endoscopic approach when jamming. However, EUS and ERCP are difficult, costly, and may be with complications. Additional operations will increase the risks and costs. Therefore, a stent that can effectively prevent reflux, solve clinical problems, and effectively prolong stent patency time is urgently needed.

DETAILED DESCRIPTION:
At present, endoscopic therapy is the preferred method to solve biliary or pancreatic diseases. And EUS-guided stent implantation and drainage of pancreatic pseudocyst is the main method in Endoscopic treatment of pancreatic pseudocyst. However, blockage of stent is a problem that has puzzled endoscopists for a long time. The mechanism of stent blockage is related to the reflux of gastrointestinal contents into the stent. Although plastic stents are widely used in patients who needed drainage. However, the average free time for stent is only 77 to 126 days, leading to the need for stent replacement in most patients within 3 months. As one end of the double pigtail stent used for drainage of pancreatic pseudocyst may be located in the stomach, it may cause the stent to be blocked by the contents of the stomach. Therefore, multiple stents or additional stents or drainage tube are often needed to further strengthen the drainage.

It seems that the mechanism of stent blockage are associated with gastrointestinal contents reflux. And stents required be replaced again by endoscopic approach when jamming. However, EUS and ERCP are difficult, costly, and may be with complications. Additional operations will increase the risks and costs. Therefore, a stent that can effectively prevent reflux, solve clinical problems, and effectively prolong stent patency time is urgently needed.

The extended enteral anti-reflux stent developed by our research team has potential advantages in prolonging the patency period of the stent and preventing secondary infection of pseudocysts. In this study, we aim to evaluate the effect of the stent on the drainage of pancreatic pseudocyst.

ELIGIBILITY:
Inclusion Criteria:

* Pancreatic pseudocyst by a variety of causes, including acute pancreatitis, chronic pancreatitis, drug-induced pancreatitis
* Pseudocyst compressed gastrointestinal or bile duct and causes obstruction symptoms or causes other symptoms
* Diameter of pseudocyst >6 cm with no compression symptoms, but progressively increases and is failed to conservatively treat

Exclusion Criteria:

* Wall-off necrosis with liquidation mimics pseudocyst
* Pseudocyst formation ≤8 weeks, cyst wall is immature
* Cannot puncture by EUS-guided approach for any reason
* Patients with serious cardiovascular or cerebrovascular diseases or other diseases which are not fitted to anaesthetize
* Severe coagulopathy or thrombocytopenia

Ages: 12 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Disappearance rate of pseudocyst（PDR） after stent implantation | in 6 months
  PDR=1-(Postoperative pseudocyst area/Preoperative pseudocyst area)×100%

SECONDARY OUTCOMES:
Time of disappearance of pseudocyst after stent implantation | in 6 months
  Time of disappearance of pseudocyst after stent implantation

CONTACTS AND LOCATIONS:
Overall Officials: Yonghui Huang, archiater, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reddy DN, Banerjee R, Choung OW. Antireflux biliary stents: are they the solution to stent occlusions? Curr Gastroenterol Rep. 2006 Apr;8(2):156-60. doi: 10.1007/s11894-006-0012-x. PMID 16533479
- [Background] Pedersen FM, Lassen AT, Schaffalitzky de Muckadell OB. Randomized trial of stent placed above and across the sphincter of Oddi in malignant bile duct obstruction. Gastrointest Endosc. 1998 Dec;48(6):574-9. doi: 10.1016/s0016-5107(98)70038-0. PMID 9852446
- [Background] van Berkel AM, Boland C, Redekop WK, Bergman JJ, Groen AK, Tytgat GN, Huibregtse K. A prospective randomized trial of Teflon versus polyethylene stents for distal malignant biliary obstruction. Endoscopy. 1998 Oct;30(8):681-6. doi: 10.1055/s-2007-1001388. PMID 9865556
- [Background] Walter D, Will U, Sanchez-Yague A, Brenke D, Hampe J, Wollny H, Lopez-Jamar JM, Jechart G, Vilmann P, Gornals JB, Ullrich S, Fahndrich M, de Tejada AH, Junquera F, Gonzalez-Huix F, Siersema PD, Vleggaar FP. A novel lumen-apposing metal stent for endoscopic ultrasound-guided drainage of pancreatic fluid collections: a prospective cohort study. Endoscopy. 2015 Jan;47(1):63-7. doi: 10.1055/s-0034-1378113. Epub 2014 Sep 30. PMID 25268308
- [Background] Aburajab M, Smith Z, Khan A, Dua K. Safety and efficacy of lumen-apposing metal stents with and without simultaneous double-pigtail plastic stents for draining pancreatic pseudocyst. Gastrointest Endosc. 2018 May;87(5):1248-1255. doi: 10.1016/j.gie.2017.11.033. Epub 2017 Dec 9. PMID 29233670
- [Background] Brimhall B, Han S, Tatman PD, Clark TJ, Wani S, Brauer B, Edmundowicz S, Wagh MS, Attwell A, Hammad H, Shah RJ. Increased Incidence of Pseudoaneurysm Bleeding With Lumen-Apposing Metal Stents Compared to Double-Pigtail Plastic Stents in Patients With Peripancreatic Fluid Collections. Clin Gastroenterol Hepatol. 2018 Sep;16(9):1521-1528. doi: 10.1016/j.cgh.2018.02.021. Epub 2018 Feb 21. PMID 29474970